CLINICAL TRIAL: NCT00255463
Title: Phase II, Placebo Controlled, Parallel Group, Double Blind, Randomised, Multicentre Trial Comparing the Anastrozole (Arimidex®) Placebo Combination to the Anastrozole - ZD1839 (Iressa™) Combination as Neoadjuvant Treatment in Postmenopausal Women With Stage I-IIIB Breast Cancer and Oestrogen Receptor (ER) and/or Progesterone (PgR) Positive Tumours
Brief Title: Phase II Neoadjuvant ER+/PgR + Arimidex +/- Iressa Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1839IL/0223; D7913C00223
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Gefitinib

INTERVENTIONS:
Drug: Anastrazole
Drug: Gefitinib

SUMMARY:
The purpose of this study is to compare the changes in a proliferation biomarker in subjects receiving Anastrozole or Anastrozole/ZD1839 combination.

ELIGIBILITY:
Inclusion Criteria:

* Measurable (stage I-IIIB) non meta static non inflammatory breast cancer
* Patients must post menopausal women who in the opinion of investigator would be likely to benefit from endocrine therapy. Postmenopausal patients are defined as:
* Natural menopause with last menses > 1 year ago,
* Radiation induced oophorectomy with last menses > 1 year ago,
* Serum FSH and LH levels clearly in the postmenopausal range for the institution.
* Bilateral oophorectomy

Exclusion Criteria:

* Other current or previous (to last 5 years) malignancies, other metastases, abnormal blood chemistry, lung/ heart/kidney/liver abnormalities,
* Hormonal treatment within the last 2 weeks, previous hormonal treatment for invasive cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 185
Dates: Start 2004-01; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
To determine and compare changes in proliferation marker at 16 weeks in the treatment groups

SECONDARY OUTCOMES:
Tumour response, safety and tolerability, pharmacokinetics, pharmacokinetics and dynamics, oestradiol levels, mastectomy rate.
Comparison of WHO and RECIST criteria,
Exploratory biomarker studies involving genomics, metabolomics and proteomics.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Iressa Medical Sciences Director, MD, Study Director — AstraZeneca
Locations (34):
- Czechia (5):
  - Research Site, Brno
  - Research Site, Chomutov
  - Research Site, Ostrava
  - Research Site, Ostrava - Poruba
  - Research Site, Prague
- France (4):
  - Research Site, Clermont-Ferrand
  - Research Site, Montpellier
  - Research Site, Tours
  - Research Site, Villejuif
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Kecskemét
- Portugal (3):
  - Research Site, Coimbra
  - Research Site, Funchal
  - Research Site, Lisbon
- Spain (6):
  - Research Site, Santiago de Compostela, A Coruña
  - Research Site, Jaén, Jaén
  - Research Site, Seville, Sevilla
  - Research Site, Valencia, Valencia
  - Research Site, Zaragoza, Zaragoza
  - Research Site, A Coruña
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Mölndal
  - Research Site, Stockholm
- United Kingdom (10):
  - Research Site, Chelmsford, Essex
  - Research Site, Bournemouth
  - Research Site, Croydon
  - Research Site, Dundee
  - Research Site, Leeds
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Poole